CLINICAL TRIAL: NCT06958185
Title: Effects of Peripheral Somatosensory Stimulation Through Mechanical Pressure on Lower Limb Muscle Strength in Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pedro Victor López Plaza (Other)
Responsible Party: Sponsor-Investigator, Pedro Victor López Plaza, Principal Investigator, Facultat de ciencies de la Salut Universitat Ramon Llull
Organization: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04-10
Record Dates: First submitted 2025-04-24; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The design of this study is a randomized crossover clinical trial. All participants (n=36) will randomly receive both the Active and Sham proprioceptive stimulation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The control group (CG) (No Intervention): The control group (CG) will have the proprioceptive stimulation device placed on the motor points of the quadriceps muscle without the application of deep sensory stimulation throughout the entire evaluation period of Maximum Strength (MS) via Mean Velocity (MV), including rest periods.
- The Experimental Group (EG1) (Experimental): The Experimental Group 1 (EG1) will have the device placed on the motor points of the quadriceps muscle with deep peripheral sensory stimulation applied via the device's plungers throughout the entire evaluation period of Maximum Strength (MS) via Mean Velocity (MV), including rest periods.
  Interventions: Device: deep peripheral sensory stimulation
- The Experimental Group (EG2) (Experimental): The Experimental Group 2 (EG2) will have the device placed on the motor points of the quadriceps muscle with deep peripheral sensory stimulation applied via the device's plungers, but only during the rest periods between repetitions in the evaluation process of Maximum Strength (MS) via Mean Velocity (MV), applied continuously for 15 seconds at 20-second intervals over a total of 5 minutes.
  Interventions: Device: deep peripheral sensory stimulation

INTERVENTIONS:
Device: deep peripheral sensory stimulation — The proprioceptive stimulus will consist of intermittent mechanical pressure on the skin, localized at the neuromuscular motor points of the rectus femoris, vastus lateralis, and vastus medialis of the quadriceps. The tissue subjected to this precise pressure in areas of high neuromuscular innervation facilitates the stimulation of kinesthetic cortical sensitivity. The experimental group (EG) will be randomly and crosswise subdivided into two groups, so that both receive the intervention in two different modalities at two different times.
  Arms: The Experimental Group (EG1); The Experimental Group (EG2)

SUMMARY:
Somatosensory information is essential for the motor system because when the central nervous system stops receiving afferent signals, it cannot use information about the state of the affected body part to plan or adjust movement. This phenomenon is known as sensory deafferentation, and it significantly affects motor function. This principle offers an opportunity to observe changes in strength through a peripheral proprioceptive stimulus that activates the muscular system with the aim of increasing recruitment. This would justify the implementation of proprioceptive input in approaches focused on motor learning in movement disorders resulting from cortical lesions such as stroke.

DETAILED DESCRIPTION:
Objective: o determine whether the application of a peripheral proprioceptive stimulus to the neuromuscular motor points of the quadriceps increases strength and muscle activation during the squat movement in the affected limb of stroke survivors.

Methods:The design of this study is a randomized crossover clinical trial. All participants (n=36) will randomly receive both the Active and Sham proprioceptive stimulation.The proprioceptive stimulus will consist of intermittent mechanical pressure on the skin, localized at the neuromuscular motor points of the rectus femoris, vastus lateralis, and vastus medialis of the quadriceps. The tissue subjected to precise pressure in these highly innervated neuromuscular zones promotes the stimulation of kinesthetic cortical sensitivity. The outcome variable will be the assessment of Maximum Strength (MS) generated by the participant during the squat movement, from a 90º knee flexion position to full extension. At the moment of peak force, the mean velocity (MV) of the concentric phase of the movement and the maximum load the participant can move will be evaluated. The intervention, assessment, and recruitment will take place at AVAN Private Foundation Sabadell and Ricard i Fortuny Socio-Healthcare Center (CSSV RiF), Vilafranca.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of unilateral hemispheric stroke (ischemic or hemorrhagic) confirmed by MRI or CT scan.
* At least 3 months must have passed since stroke onset.
* Ability to stand independently in a static position or to walk, regardless of whether assistance is needed.

Exclusion Criteria:

* Diagnosis of cognitive, visual, or cardiorespiratory disorder (including the presence of a cardiac pacemaker, heart failure, arrhythmia, or severe COPD)
* Orthopedic intervention in the lower limb
* Balance disorders of vestibular origin
* Skin diseases
* Botulinum toxin treatment within the past year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Strength (MS) | estimated time of movement and data collection of 20 minutes
  The outcome variable will consist of the assessment of Maximum Strength (MS) generated by the participant during the squat movement, from a 90º knee flexion position to full extension measured in two units, kilograms and newtons.

OTHER OUTCOMES:
electric neuromuscular activation electric neuromuscular activation electric neuromuscular activation | estimated time of movement and data collection of 20 minutes
  In addition to strength assessment, portable sensors will be placed to digitize the electrical activity (surface electromyography), related to the variable of neuromuscular activation during the squat movement.
Transfer of body weight support onto the affected limb in relation to the unaffected limb | estimated time of movement and data collection of 20 minutes
  Pressure insoles, one on each foot, to record plantar pressure distribution and obtain ground reaction forces.

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Victor López Plaza, Barcelona, Spain